CLINICAL TRIAL: NCT00166725
Title: A Randomized, Open Label, Multicenter Study Evaluating the Effects of Octreotide Acetate on Circulating Levels of Chromogranin A in Advanced Prostate Cancer Patients
Brief Title: Effects of Octreotide Acetate on Circulating Levels of Chromogranin A in Advanced Prostate Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSMS995A2402
Record Dates: First submitted 2005-09-07; First posted 2005-09-14 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Prostate Cancer
Keywords: HRPC; octreotide LAR; CgA
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Drug: Octreotide LAR

SUMMARY:
The present study will provide information on whether the somatostatin analog, octreotide acetate, could have an inhibitory effect on circulating chromogranin A. The demonstration of an antisecretory effect of somatostatin analogs could offer a rationale for a large scale randomized study.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients aged >18
2. ECOG performance status < 3
3. Patients with metastatic prostate cancer currently receiving 1st line hormonal therapy (LHRH agonists or surgical castration) and failing with raising serum PSA
4. Biochemical progression documented by three consecutively rising serum PSA measurements, each separated from the other by at least 2 weeks, with the last measurement being 50% or greater than the nadir PSA achieved after the last therapeutic maneuver (i.e. first line hormonal therapy noted above)
5. Demonstrated tolerance to a test dose of s.c. octreotide acetate injection at Visit 1
6. Elevated (> 40 U/L according to DAKO Elisa kit) chromogranin A plasma levels documented by at least two consecutive measurements
7. Liver function tests < 2.5 ULN, serum creatinine within normality
8. Serum PSA (50% increased value) above 4 ng/mL for patients with intact prostate and > 0.8 ng/mL for post prostatectomy patients at study entry
9. Immediate history of rising PSA < 10 months
10. Castrate levels of testosterone (< 30 ng/dL)
11. Life expectancy of > 6 months
12. Signed informed consent prior to initiation of any procedure

Exclusion Criteria:

1. Prior chemotherapy or other systemic anticancer therapy except for LHRH agonists, and/or non-steroidal anti-androgens (eg, flutamide, bicalutamide or nilandron)
2. Palliative radiotherapy less than 6 weeks (42 days) prior to planned entry date
3. Other investigational drugs within the past 28 days
4. Long-term (> 3 months) treatment with proton pump inhibitors
5. Uncontrolled blood hypertension
6. Other malignancies within 5 years prior to study entry, except for curatively treated non-melanotic skin cancer
7. Patients with another non-malignant disease which would confound the evaluation of the primary endpoints or prevent the patient from complying with the protocol

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-02

PRIMARY OUTCOMES:
Time to 25% decrease in chromogranin A plasma level (evaluation every 4 weeks for the first 12 weeks and every 12 weeks after)

SECONDARY OUTCOMES:
PSA response (decrease > 50% or increase > 25% from baseline)
Time to symptomatic progression (bone pain increase, deterioration of ECOG performance status)
Change in circulating IGF-1, VEGF, IL-6, serum alkaline phosphatase, serum creatinine and serum calcium every 4 weeks for the first 12 weeks and every 12 weeks after

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Orbassano, Orbassano, Italy